CLINICAL TRIAL: NCT06936319
Title: Physical Counterpressure Maneuvers in Postural Orthostatic Tachycardia Syndrome (POTS) - a Monocentric, Randomized Controlled Trial
Brief Title: Counterpressure Maneuvers in Postural Orthostatic Tachycardia Syndrome
Acronym: CPM_in_POTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20241114-3611
Record Dates: First submitted 2025-03-28; First posted 2025-04-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-03

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS)
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best clinical practice (Active Comparator): Counselling on counterpressure maneuvers and other behavioral and non-pharmacological measures to combat POTS symptoms in daily life.
  Interventions: Other: Best clinical practice
- Best clinical practice plus CPM-biofeedback training (Experimental): In addition to counselling on CPM and other behavioral and non-pharmacological measures to combat POTS symptoms in daily life, participants undergo a CPM-biofeedback training session in the autonomic function laboratory under continuous HR and BP monitoring.
  Interventions: Behavioral: Best clinical practice plus CPM-biofeedback training

INTERVENTIONS:
Behavioral: Best clinical practice plus CPM-biofeedback training — The CPM-biofeedback training consists of a baseline 2-minutes active standing and the following four different physical maneuver: leg crossing and muscle tensing, heel raises (10 tiptoeing per minute), squatting, unilateral handgrip (20 times per minute). All exercises will be performed under continuous heart rate and blood pressure monitoring to enable the study participants to gain feedbacks on the effect of the maneuvers on their own biosignals.
  Arms: Best clinical practice plus CPM-biofeedback training
Other: Best clinical practice — Recommendations about life-style and behavioural measures to mitigate POTS symptoms in daily life.
  Arms: Best clinical practice

SUMMARY:
The present study evaluates whether performing a 14-days counter pressure maneuvers (CPM)-biofeedback training improves the symptomatic burden (primary objective) and secondarily the interference of POTS symptoms with daily activities, fatigue, and health-related quality of life of individuals with POTS compared to best clinical practice non-pharmacological measures. Secondary in-laboratory objectives are to assess the influence of CPM on the supine-to-standing heart rate (HR) and blood pressure (BP) changes as well as on the severity of orthostatic intolerance after performing CPM for two minutes compared to a baseline (intervention-free) active standing test, and to assess the safety and tolerability of CPM-biofeedback training in individuals with POTS.

This is a monocentric, proof-of-concept, 1:1 randomized, controlled trial with rater-blinded evaluation of the hemodynamic effect of CPM in 40 individuals suffering from POTS.

All study participants will receive detailed counselling on CPM and other behavioral and non-pharmacological measures to combat POTS symptoms in daily life and will be invited to practice them regularly (best clinical practice). Participants randomized to the interventional arm will receive a CPM-biofeedback training session in the autonomic function laboratory at the Department of Neurology of the Innsbruck Medical University to learn four different CPM under continuous HR and BP monitoring. The CPM-biofeedback training will consist of a baseline 2-minutes active standing and the following four different physical maneuver: leg crossing and muscle tensing, heel raises (10 tiptoeing per minute), squatting, unilateral handgrip (20 times a minute).

The trial foresees three study visits for both the interventional and the control arm (screening and baseline on-site, as well as a telephone visit 14 days later). For the interventional trial arm, two additional visits are planned (CPM-biofeedback training session in the autonomic function laboratory and a follow-up telephone visit 7 days later).

To evaluate the baseline to day-14 change in symptom severity, the Malmö POTS Score (MAPS) total score (primary endpoint) and the MAPS single items, Vanderbilt Orthostatic Symptom Score, Orthostatic Grading Scale, Fatigue Severity Scale and Health-related Quality of Life Questionnaire (EuroQol -EQ-5D-5L ) will be administered.

ELIGIBILITY:
Inclusion Criteria:

* POTS diagnosis
* 18 to 80 years of age at time of consent
* stable medication in the seven days prior to the baseline visit
* able to provide written informed consent

Exclusion Criteria:

* participation in other interventional trials
* pregnant or breastfeeding females
* on treatment with vasoactive medications including medications for heart rate control
* acute infections at the time of enrolment or in the two weeks before
* acute pain
* surgery in the last three months
* inability or contraindication for performing hip and knee flexion, hip adduction or squatting
* inability to stand for at least two minutes
* Any other cardiological, internal, psychiatric or neurological condition, which may prevent engagement in the sturdy procedures in the judgement of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Malmö Postural Orthostatic Tachycardia Syndrome symptom score (MAPS) | Baseline to day-14
  Baseline to day-14 change in the total score from 0 to 120. Higher scores means more symptoms and higher symptom severity.

SECONDARY OUTCOMES:
Severity of orthostatic intolerance (on a 0 - 10 points scale) | After performing four different counterpressure maneuvers for two minutes each during the biofeedback session, at day 1 +/-3.
  Secondary in-laboratory endpoint, orthostatic intolerance after two minutes upon standing and performing counterpressure maneuvers compared to a baseline active standing for two minutes; higher score means more severe symptoms of orthostatic intolerance.
Absolute heart rate | At 15, 30, 60, 90 and 120 seconds during four different counterpressure maneuver practiced upon standing , at day 1 +/-3.
  Absolute heart rate compared to baseline active standing.
Absolute systolic and diastolic blood pressure | At 15, 30, 60, 90 and 120 seconds during counterpressure maneuver practiced upon standing, , at day 1 +/-3.
  Absolute systolic and diastolic blood pressure at 15, 30, 60, 90 and 120 seconds during counterpressure maneuver practiced upon standing compared to baseline active standing.
Supine-to-standing change in heart rate | At 15, 30, 60, 90 and 120 seconds during four different counterpressure maneuvers, at day 1 +/-3.
  Supine-to-standing change in heart rate at 15, 30, 60, 90 and 120 seconds during four different counterpressure maneuver compared to baseline active standing (same timepoints)
Supine-to-standing change in systolic and diastolic blood pressure | At 15, 30, 60, 90 and 120 seconds during four different counterpressure maneuvers, at day 1 +/-3.
  Supine-to-standing change in systolic and diastolic blood pressure compared to baseline active standing at 15, 30, 60, 90 and 120 seconds during four different counterpressure maneuvers
Single items of the Malmö POTS Score (MAPS) | Baseline to day-14
  Baseline to day-14 change in twelve single items of the Malmö POTS Score (MAPS) from 0-10. Higher scores indicate more severe symptoms.
Vanderbilt Orthostatic Symptom Score (VOSS) | Baseline to day-14
  Baseline to day-14 change in the 9 items Vanderbilt Orthostatic Symptom Score (VOSS, score range: 0-90). A higher score means more pronounced symptoms.
Orthostatic Grading Scale (OGS) | Baseline to day-14
  Baseline to day-14 change in the 5-items Orthostatic Grading Scale (OGS, score range: 0-20). Higher scores mean more interference of daily life due to symptoms.
Fatigue Severity Scale (FSS) - german Version | Baseline to day-14
  Baseline to day-14 change in the 9-items Fatigue Severity Scale (FSS) - german Version (score range: 1 to 63). Higher scores mean pronounced symptoms and worse outcome.
European Quality of Life, 5 Dimensions, 5 Levels (EuroQol -EQ-5D-5L - german Version) | Baseline to day-14
  Baseline to day-14 change in the 5-items EuroQol -EQ-5D-5L - german Version and a 0-100 visual analogue scale. Higher scores means better outcome and self-estimated health, 100= best, 0= worse health.
Estimated number and preferred choice of counterpressure maneuvers in daily life | Baseline to day-14
  Baseline to day-14 estimated number and preferred choice of counterpressure maneuver in daily life. Higher numbers indicate that a given counterpressure maneouver was performed more frequently, and stand for a better compliance.
Overall usefulness of counterpressure maneuvers | Baseline to day-14
  Overall usefulness of counterpressure maneuvers on a Likert scale 0-10. Higher scores indicate higher subjective usefulness of a given counterpressure maneouver.
Adverse events | Screening-Visit to day-14
  Any adverse event from screening to day-14.
Barriers to counterpressure maneuver application in daily life | Baseline to day-14
  Barriers to counterpressure maneuver application in daily life in the opinion of the study participants. Open answers possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided